CLINICAL TRIAL: NCT06029218
Title: Analysis of the Toxicity and Efficacy of Daily 1 vs 2 Beam Proton Therapy : Analysis of the Toxicity and Efficacy of Daily 1 vs 2 Beam Proton Therapy
Brief Title: Analysis of the Toxicity and Efficacy of Daily 1 vs 2 Beam Proton Therapy
Acronym: P1V2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/72
Record Dates: First submitted 2023-07-25; First posted 2023-09-08 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Chordoma; Chondrosarcoma; Ewing Sarcoma; Osteosarcoma
Keywords: protontherapy
MeSH Terms: conditions — Chordoma; Chondrosarcoma; Sarcoma, Ewing; Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1DB (Experimental): One daily Beam treatment
  Interventions: Radiation: Proteus ONE one daily beam
- 2DB (Active Comparator): Two daily beam goldstandard
  Interventions: Radiation: Proteus ONE two daily beam

INTERVENTIONS:
Radiation: Proteus ONE one daily beam — A single daily beam is used, doubling the dose delivered for this treatment incidence.
  Arms: 1DB
Radiation: Proteus ONE two daily beam — two daily beams are used, in accordance with the initial treatment plan and the patient's standard of care
  Arms: 2DB

SUMMARY:
Thanks to the intrinsic qualities of the proton beam, proton therapy will reduce adverse effects of irradiation. The Proteus®One is the latest generation of proton therapy equipment, enabling the Centre Antoine Lacassagne to expand its range of treatments by carrying out new proton therapy treatments. It has an innovative compact isocentric rotating head (Gantry) that allows the radiation beam to be directed at different angles around the patient. In some cases, two beams are used to treat tumours, and by convention, both beams are delivered during the same session. However, it is necessary to position the patient before each beam, which is time-consuming because 2 beams have to be positioned very precisely each day. The aim of this study is therefore to assess the toxicity of proton therapy delivered by a single daily beam compared with proton therapy delivered by two daily beams, which is the conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* Chordoma, chondrosarcoma of the skull base and spine, Ewing's sarcoma, and osteosarcoma meeting the criteria for treatment by proton therapy
* Tumour requiring 2 beams
* MRI less than one month old
* PS 0-2.
* Patient who has read the patient information note and signed the consent form.
* Patient with healthcare insurance cover.
* Age over 18 years.
* For women of childbearing age, negative urine pregnancy test and effective contraception in place for the duration of treatment and for six months following the end of treatment.

Exclusion Criteria:

* Persons deprived of their liberty or under guardianship.
* Unable to undergo the medical follow-up of the clinical investigation for geographical, social or psychological reasons.
* Patient eligible for symptom reduction surgery Vulnerable populations and participants defined in Articles 64 to 68 of Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the frequency of occurrence of toxicities in the group of patients treated with two daily beams (2DB) and in the group of patients treated with one daily beams (1DB). | During 2 to 7 weeks of protontherapy treatment and during 5 years follow-up
  Assessment of the incidence of grade ≥2 medical device-related toxicities assessed according to CTCAE version 5.0 in each of the two treatment arms.

SECONDARY OUTCOMES:
Determining the effectiveness of proton therapy | 5-year follow-up visits
  Efficacy will be assessed in terms of relapse rate
Determining the effectiveness of proton therapy | 5-year follow-up visits
  Efficacy will be assessed in terms of local control by MRI assessment
Determining the effectiveness of proton therapy | 5 years follow-up
  Efficacy will be assessed in terms of overall survival
Quality of life assessment | During 2-7 weeks of protontherapy treatment and during 5 years follow-up
  Quality of life will be assessed using the EORTC QLQ-C30 scale (Appendix 2), version 3 at the inclusion assessment, at the end-of-treatment visit and at each assessment visit for five years. Version 3.0 of the QLQ-C30 has four-point scales for the items 1 to 28 namely : 1 : "Not a tall", 2 : "A little", 3 : "Quite a bit" and 4 : "Very much." Higher score mean worse outcome. Item 29 and 30 has seven-point scales from 1 : " very bad " to 7 "Excellent". Lower score mean worse outcome.
Evaluate the time saving between the two arms 1DB and 2DB | 2-7 weeks of protontherapy treatment
  Time savings will be assessed by measuring the time taken for door-to-door proton therapy treatment sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No